CLINICAL TRIAL: NCT01760642
Title: Identification and Evaluation of Endogenous Markers for the Assessment of CYP3A Activity in Female Subjects Using Metabolomics
Brief Title: Identification and Evaluation of Endogenous Markers for the Assessment of CYP3A Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joo-Youn Cho, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYP_metabolomics
Record Dates: First submitted 2012-12-26; First posted 2013-01-04 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: metabolite profiles; pharmacokinetics; CYP3A; metabolomics
MeSH Terms: interventions — Midazolam; Long-Term Synaptic Depression; Ketoconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midazolam (Experimental): period 1: midazolam 1 mg IV single dose administration. period 2: midazolam 1 mg IV single dose after ketoconazole 400 mg oral dosing for 3 days.
  period 3: midazolam 2.5 mg IV single dose after rifampicin 600 mg oral dosing for 10 days.
  Interventions: Drug: Midazolam; Drug: Ketoconazole; Drug: Rifampicin

INTERVENTIONS:
Drug: Midazolam — Midazolam 3 mg IV
  Other Names: Midazolam (Bukwang Pharm.Co., Ltd.)
Drug: Ketoconazole — ketoconazole 400 mg PO
  Other Names: Kaszole (Skynewpharm Inc.)
Drug: Rifampicin — Rifampicin 600 mg PO
  Other Names: Rifampin (Yuhan Corp.)

SUMMARY:
Identification and evaluation of endogenous markers for the assessment of CYP3A activity in female subjects using metabolomics

DETAILED DESCRIPTION:
Eligibility for participation of this study will be determined from demographic information, medical history, physical examination, electrocardiogram(ECG) and clinical laboratory tests within 3 weeks before study drug administration. Subjects suitable for this study will be admitted to the Clinical Trials Center, Seoul National University Hospital on the day before dosing, and they will be overnight-fasted from 9 p.m. of Day -1. Urine collection is scheduled from 24 hours before midazolam administration to 24 hours after administration. Subjects will be dosed midazolam by intravenous around at 9 a.m. of Day 1. Subjects will perform scheduled procedures including clinical laboratory tests, electrocardiograms and pharmacokinetic samplings. Subjects will be discharged on Day 2 and visit the Clinical Trials Center for period 2, ketoconazole administration. After 3 days of ketoconazole administration, midazolam will be dosed with ketoconazole on Day 4 of period 2. Subjects will perform scheduled procedure and on period 3 rifampicin will be dosed for 9 days and on Day 10 of period 3 midazolam will be dosed with rifampicin. After subjects perform scheduled procedure, the study will be terminated 6-8 days after the end of period 3.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 50 years of age, inclusive
* Weight: Between 45 to 95 kg, within 17 - 28 of Body Mass Index
* Menstruation cycle between 21 to 35 without contraceptive
* Subject who agree contraception during the study
* Subject who are reliable and willing to make themselves available during the study period, are willing to follow the study protocol, and give their written informed consent voluntarily

Exclusion Criteria:

* History of hypersensitive reaction to medication (midazolam, ketoconazole, rifampicin)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease history or evidence of drug abuse
* A subject whose lab test results are as follows; Liver function test (AST, ALT, GGT, ALP, LDH, Total bilirubin) > 1.25 X upper limit of reference range
* A subject whose SBP is over 140 mmHg or below 90 mmHg and DBP is over 100 mmHg or below 50 mmHg
* Presence or history of drug abuse or positive result in urine drug screening test
* Blood donation during 2 months or apheresis during 1 month before the study
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any OTC medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
* Use of alcohol over 21 units/weeks
* Smoker who smoke more than 10 cigarettes per day
* Participation in clinical trials of any drug within 60 days prior to the participation of the study
* Use of grapefruit juice within 1 week before first dose
* Use of caffeine drink within 3 days before first dose
* Subject pregnant or breast-feeding
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Metabolomic profile | -24--12h, -12-0h of every midazolam dosing
  endogenous metabolite profiles such as steroid

SECONDARY OUTCOMES:
Pharmacokinetics | 0h, 10m, 20m, 30m, 45m, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h of every midazolam dosing
  Cmax, AUClast of midazolam

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Youn Cho, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National Universtiy Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin KH, Ahn LY, Choi MH, Moon JY, Lee J, Jang IJ, Yu KS, Cho JY. Urinary 6beta-Hydroxycortisol/Cortisol Ratio Most Highly Correlates With Midazolam Clearance Under Hepatic CYP3A Inhibition and Induction in Females: A Pharmacometabolomics Approach. AAPS J. 2016 Sep;18(5):1254-1261. doi: 10.1208/s12248-016-9941-y. Epub 2016 Jun 17. PMID 27317471